CLINICAL TRIAL: NCT06522191
Title: Effect of Cross Education Using Robotic Rehabilitation on Upper Extremity Motor Function and Strength in Stroke Patients
Brief Title: Cross Education for Upper Extremity Motor Function and Strength in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Rüstem Mustafaoğlu, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/83
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Cross education; Cross training; Robotic rehabilitation; Upper extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cross-Education (CE) Group (Experimental): Participants in the CE group will receive repetitive task practice through a robotic rehabilitation (RR) device on the less-affected upper extremity for 20 minutes, twice a week, for 5 weeks, in addition to a physical therapy (PT) program provided 5 days a week. This CE training will be conducted prior to the RR sessions performed on the more affected UE within the PT intervention to facilitate cross-education and support motor priming. In this study, RR applications will utilize an intelligent feedback RR system.
  Interventions: Other: Physiotherapy Training (PT); Device: Cross-Education Intervention
- Control Group (Sham Comparator): Participants in the control group will be given lower extremity-focused exercises for 20 minutes, twice a week, for 5 weeks before the RR application included in the PT program, in order to eliminate the potential effect of the additional treatment provided in the study.
  Interventions: Other: Physiotherapy Training (PT); Other: Control Intervention

INTERVENTIONS:
Other: Physiotherapy Training (PT) — Both groups received the same therapist-led standardized PT for 5 days a week including 2 days of RR plus 3 days of conventional rehabilitation (CR) for 5 weeks. RR training will be given 40 min per session using an intelligent feedback robotic system. The system allows patients to move a cursor to targets on a monitor using a unilateral exoskeleton robotic arm and handle, which supports shoulder, elbow, forearm, and optionally multi-joint movements. The system provides visual and auditory feedback, offering exergame training with 1Dimension (D), 2D, and 3D options adjustable to three levels (low to high). Exergames and their parameters will be customized based on each patient's capacity. The CR protocol consists of joint range-of-motion, correct movement, stretching and balance exercises, gait training (walking on level surfaces, stairs), strengthening of antagonist muscle pattern will be provided. Each CR session will last 45 min of active treatment.
Device: Cross-Education Intervention — Participants in the CE group will have the less affected upper extremity undergo game-based, unilateral, repetitive movement training using RR to enhance the effectiveness of the training to be provided to the affected side. Similar therapeutic games (exergames) planned for the more affected upper extremity will be selected through the unilateral exoskeleton RR device. As described in the PT section, upper extremity movements will be performed using the robotic arm and handle during the games. The difficulty level will be adjusted by the supervisor physiotherapist based on the grip threshold on the robotic handle, the game's difficulty level (low to high), workspace arrangement before each session, and suspension level according to the patient's needs. An approximately 20-minute program will be implemented, consisting of 8 games, each lasting about 2.5 minutes, tailored to the patient's capacity.
  Arms: Cross-Education (CE) Group
Other: Control Intervention — The exercises to be administered in the control intervention will be selected based on the patient's level of impairment but will be planned without progression or intensity increase, and the involvement of the upper extremity will be kept to a minimum. The exercises will include lower limb joint range of motion exercises, weight bearing, weight shifting, and gait training.
  Arms: Control Group

SUMMARY:
Stroke is the leading cause of disability and mortality worldwide. The impact of stroke on the upper extremity functions is a common and important cause of long-term disability. Indeed, six months after the stroke, a considerable amount of patients are still unable to incorporate the affected upper limb into their daily activities. On the other hand, weaknesses are also observed in the "apparently normal" ipsilateral side of the lesion due to the presence of corticospinal fibers that do not cross to the contralateral side of the medulla.

This study aims to investigate the effects of cross-education (CE) using robotic rehabilitation on upper extremity motor function and strength in patients with stroke. Secondary objectives include assessing quality of life and activities of daily living.

Researchers will compare CE using robotic rehabilitation to the control group (CON) that received lower extremity-focused exercises to see if CE works to enhance rehabilitation outcomes.

Participants will receive 20 min, twice weekly CE (to the less affected upper limb) or CON before the RR intervention included in the PT intervention administered 5 days in a week for 5 weeks. They will be evaluated using the relevant outcomes at the beginning and the end of the study (5th week).

DETAILED DESCRIPTION:
After a stroke, upper extremity strength and skill deficits are predominant on the paretic side. In the chronic phase of stroke, patients with moderate to severe impairment also experience functional deficits on the less affected side, increasing dependence on this extremity during daily living activities. This situation highlights the necessity of incorporating the non-affected side into rehabilitation. Current rehabilitation approaches focus on intensive, highly repetitive, and task-oriented training. The aim within this framework is to induce neuroplasticity in the lesioned hemisphere to promote motor recovery. Techniques such as constraint-induced movement therapy are effective for inducing neuroplastic changes but are not suitable for all patient populations. Therefore, alternative treatment strategies are needed to induce neuroplastic changes in patients with greater upper extremity disability.

As stated above, promoting lesional hemispheric reorganization is crucial for recovery; however, the role of the contralesional motor cortex in recovery remains debated. Rehabilitation strategies must be tailored to the severity of motor impairment in patients. Cross-education (CE) emerges as a novel alternative rehabilitation strategy for individuals with moderate to severe motor impairment on the affected side. CE refers to the improvement in strength or skill in the contralateral limb through unilateral motor training. For stroke patients, this can be defined as gains in the paretic extremity through the training of the less affected side. Two main hypotheses underlie CE: the "cross-activation" and "bilateral access". The cross-activation model posits that unilateral activity stimulates both ipsilateral and contralateral cortical motor areas, whereas the bilateral access model suggests that training one side leads to adaptation in the untrained muscle on the opposite side via communication between motor areas in both hemispheres. Evidence indicates that in stroke patients, the corticospinal excitability of the affected hemisphere increases with CE-induced gains. functional magnetic resonance imaging (fMRI) studies in healthy individuals show that CE results in expanded activation areas in the contralateral sensorimotor cortex and the ipsilesional temporal lobe.

To date, studies on stroke involving CE have included strengthening exercises and task-oriented functional skill training, appearing effective in improving motor function and strength. Studies have shown that strength gains in stroke patients are greater compared to neurologically intact individuals. Robotic rehabilitation has proven effective in improving upper extremity motor functions and strength in stroke patients. However, no studies have investigated CE provided through unilateral robotic rehabilitation. This study aims to evaluate the effect of CE provided by an exoskeleton-type unilateral upper extremity robotic rehabilitation device on upper extremity motor function and strength.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke more than 3 months of stroke onset
* History of first-ever unilateral ischemic or hemorrhagic stroke
* Upper extremity motor impairment; defined by an upper extremity score ≤42 on the Fugl Meyer upper extremity (FM-UE) assessment.
* No excessive spasticity in the affected arm (Modified Ashworth Scale ≤3)
* Having the ability to communicate and understand instructions (Mini-mental state examination ≥ 24)
* Being able to sit without needing any additional support and without leaning on a backrest

Exclusion Criteria:

* Cardiovascular instability (severe, uncontrolled hypertension, coronary artery disease, etc.)
* Other neurological or musculoskeletal problems that can affect upper extremity functions
* Severe upper extremity pain defined as >7 on the Visual Analogue Scale
* Botox injections of the upper extremity within 3 months before enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Change Score of Fugl-Meyer Assessment - Upper Extremity (FM-UE) | Baseline, post-intervention (approximately 5 weeks)
  We will use the upper extremity subscale of the Fugl-Meyer Assessment (FM-UE), a scale sensitive to therapeutic changes in the post-stroke period, to evaluate motor impairment. The FM-UE assesses movements and reflexes of the shoulder, elbow, forearm, wrist, fingers, ranging from proximal to distal and from synergistic to isolated voluntary movements. There are 33 upper extremity items, and the score ranges from 0 to 66, with higher scores indicating better performance. Each item in the FM-UE is rated on a 3-point ordinal scale (0= cannot perform, 1= performs partially, 2= performs fully). The FM-UE has excellent reliability and validity in stroke patients.
Change Score of Action Research Arm Test (ARAT) | Baseline, post-intervention (approximately 5 weeks)
  Upper extremity motor function will be measured by the ARAT. It includes 19 items divided into four subscales (grasp, grip, pinch, and gross movement subscales) that encompass the main aspects of arm and hand use in daily activities, with a total score ranging from 0 to 57, where higher scores indicate better performance. Most items evaluate the ability to grasp objects of different shapes and sizes and move them to various vertical or horizontal positions. Each item is scored on a 4-point scale (0: cannot perform any part of the task; 1: performs the task partially; 2: completes the task but with abnormal movement components or body posture, or the task takes more than 5 seconds but less than 1 minute to complete; 3: completes the task normally within the 5-second time limit). During the assessment, the time taken for the patient to complete each task will be measured using a stopwatch, and the patient will be observed throughout the task to assign a score based on their performance.
Change Score of Box and Block Test (BBT) | Baseline, post-intervention (approximately 5 weeks)
  The BBT test will be used to measure unilateral gross manual dexterity. It primarily evaluates gross motor function. There are 150 piece 2.5 cm³ blocks in a test box. The patient will be asked to grasp as many cube blocks as possible from the compartment of the side being tested and transfer them one by one over a barrier to the other compartment (horizontal adduction) within one minute. The instruction given to patients is: "I want to see how quickly you can pick up a block with your right (or left) hand and transfer it to the other side, one at a time". The score of the test is determined by the number of blocks correctly transferred to the other compartment within one minute.
Change Score of Isometric Grip Strength | Baseline, post-intervention (approximately 5 weeks)
  The isometric hand grip strength of both sides will be measured using a hydraulic hand dynamometer. The participant will be asked to squeeze the dynamometer for a trial attempt. When the participant is ready, they will squeeze the dynamometer with maximum isometric contraction for 5 seconds. The participant should be encouraged to exert maximum effort. The purpose of the trial attempt is to ensure that the participant understands the procedure. After the trial attempt, the participant will be instructed to squeeze as hard as possible. Both sides will be evaluated three times with one-minute rest intervals between each attempt, and the average of the three measurements will be taken. The patient will be in a seated position with the shoulder adducted, elbow flexed at 90°, forearm, and wrist in a neutral position. Support against gravity will be provided as needed to maintain the position.
Change Score of Isometric Muscle Strength | Baseline, post-intervention (approximately 5 weeks)
  To evaluate the maximum isometric muscle strength of the elbow flexors and extensors on both sides, a Lafayette hand dynamometer (Model 01163, Lafayette Instrument Co, Lafayette, Indiana) will be used. In the study, for the assessment of elbow flexor and extensor muscle strength, the patient will be positioned supine with the shoulder, forearm, and wrist in a neutral position (0°), the elbow at 90° flexion, and the fingers in a flexed position. The dynamometer pads will be placed and secured proximally on the radial and ulnar styloid processes to measure elbow flexion and extension strength, respectively. Continuous verbal encouragement will be provided during the test. Patients will be asked to perform a maximum isometric contraction, and a submaximal contraction will be performed before the evaluation to prepare for the assessment. A total of three assessments will be conducted with 30-second rest intervals, and the average of the data (in kg) will be recorded.

SECONDARY OUTCOMES:
Change Score of Stroke Impact Scale (SIS) | Baseline, post-intervention (approximately 5 weeks)
  The Turkish version of the SIS 3.0 will be used to evaluate function and health-related quality of life (HRQoL). The questions are based on subjective reports across eight clinically relevant domains. It consists of two parts. The first part is the primary scale of the SIS, which evaluates multidimensional HRQoL, including strength, hand function, activities of daily living (ADL)/ instrumental ADL, mobility, communication, emotion, memory/thinking, and social participation. It comprises 59 items, each scored using a 5-point Likert scale based on the difficulty perceived over the past week. The second part of the SIS includes an assessment of stroke recovery using a scale ranging from 0 to 100 (0: no recovery, 100: full recovery). Each domain score is converted to a score out of 100, and the mean scores of all domains are used to represent the HRQoL. The formula used for converting each domain score is 'Domain Score = [(actual - possible raw score) / possible raw score range] x 100'.
Change Score of Barthel Index (BI) | Baseline, post-intervention (approximately 5 weeks)
  The level of independence in patients' activities of daily living will be determined by the Barthel Index (BI). It consists of ten items assessing mobility and self-care activities of daily living. The scoring range is from 0 to 100; a score range of 0 to 20 represents total dependency; 21 to 61 indicates severe dependency; 62 to 90 indicates moderate dependency; 91 to 99 indicates mild dependency, and a score of 100 represents complete independence.
Adverse Events | Any adverse event reported during the 5 weeks of intervention protocol.
  Any adverse event or near miss is required to be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Aykut CAVDAR, BSc, Principal Investigator — Istanbul University-Cerrahpasa, Institute of Graduate Studies, Department of Physiotherapy and Rehabilitation; Rustem MUSTAFAOGLU, PhD, Study Chair — Istanbul University-Cerrahpasa, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation; Belgin ERHAN, PhD, Study Director — Physical Medicine and Rehabilitation Department, Faculty of Medicine, Istanbul Medeniyet University
Locations (1):
- Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoykov ME, Corcos DM, Madhavan S. Movement-Based Priming: Clinical Applications and Neural Mechanisms. J Mot Behav. 2017 Jan-Feb;49(1):88-97. doi: 10.1080/00222895.2016.1250716. Epub 2017 Mar 1. PMID 28277966
- [Background] Lim H, Madhavan S. Effects of Cross-Education on Neural Adaptations Following Non-Paretic Limb Training in Stroke: A Scoping Review with Implications for Neurorehabilitation. J Mot Behav. 2023;55(1):111-124. doi: 10.1080/00222895.2022.2106935. Epub 2022 Aug 8. PMID 35940590